CLINICAL TRIAL: NCT02712047
Title: A Randomised, Placebo-controlled, Double-blind, Two Period Crossover Study to Characterise the Exhaled Nitric Oxide Time Profile as a Biomarker of Airway Inflammation in Adult Asthma Patients Following Repeat Administration of Inhaled Fluticasone Furoate (FF)/ Vilanterol (VI) 100/25 mcg.
Brief Title: A Phase IIA FF/VI Study to Measure FeNO in Asthmatic Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201499
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: Fluticasone furoate/vilanterol; Asthma; fraction of exhaled nitric oxide; cross-over
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluticasone furoate/vilanterol (FF/VI) 100/25 mcg (Experimental): Subjects will receive FF/VI 100/25 mcg each morning (once daily) from Day 1 to Day 14, followed by a 21-day monitoring/washout period
  Interventions: Drug: Fluticasone furoate (FF) (100 mcg); Drug: Vilanterol (VI) (25 mcg)
- Placebo (Placebo Comparator): Subjects will receive placebo each morning (once daily) from Day 1 to Day 14, followed by a 21-day monitoring/washout period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone furoate (FF) (100 mcg) — First blister strip contains FF blended with lactose, 100 mcg per blister
  Arms: Fluticasone furoate/vilanterol (FF/VI) 100/25 mcg
Drug: Vilanterol (VI) (25 mcg) — Second blister strip contains vilanterol blended with lactose and magnesium stearate, 25 mcg per blister
  Arms: Fluticasone furoate/vilanterol (FF/VI) 100/25 mcg
Drug: Placebo — Matching placebo will have two blister strips, identical in appearance to the inhaler containing active study medication; one containing lactose and the second strip containing lactose and magnesium stearate
  Arms: Placebo

SUMMARY:
For asthmatic subjects, a combination of inhaled corticosteroid (FF) and long-acting beta2 receptor agonist (VI) is recommended for use (once daily) and fraction of exhaled nitric oxide (FeNO) is a non-invasive airway inflammation marker.

In this randomised, double blind, placebo-controlled, two-period, crossover repeat dose study, the duration of action of fluticasone furoate (FF) will be determined by monitoring the return of FeNO levels to baseline, following the treatment with FF/vilanetrol (VI) in asthmatic subjects.

Subjects who meet the eligibility criteria will participate in the following two treatment periods: FF/VI 100/25 mcg once-daily and placebo once-daily. Approximately 28 subjects will be enrolled in order to achieve 24 evaluable subjects. A 2-week treatment period will be followed by a 21-day monitoring/washout period before crossing over to the next treatment period. Total duration of each subject will be a maximum of 21 weeks. FeNO will be monitored up to 21 days after treatment with FF/VI together with FEV1 (up to 7 days).

ELIGIBILITY:
Inclusion Criteria:

* Age of subject: Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A doctor diagnosis of asthma for at least 6 months prior to the start of the study.
* Severity of disease: A screening pre-bronchodilator forced expiratory volume in one second (FEV1) >=60% of predicted values, which will be based upon NHANES III
* Reversibility of disease: Demonstrated presence of reversible airway disease at screening (repeat testing of eligibility can be undertaken following the screening visit up to Day -7) OR The presence of reversible airways disease can have been demonstrated historically within 6 months of the screening visit. Reversible airway disease is defined as increase in FEV1 of >=12% over baseline and an absolute change of >=200 mL within 30 minutes following 4 inhalations of albuterol/salbutamol inhalation aerosol/spacer (or equivalent nebulised treatment with albuterol/salbutamol solution).
* Current Therapy: Short-acting beta2-agonists (SABA) prescribed for at least 12 weeks prior to screening. No inhaled corticosteroids (ICS), long-actint beta2-receptor agonist (LABA), long acting muscarinic anatagonist (LAMA), leukotriene receptor antagonist (LTRA) therapy for three months prior to the start of the study.
* Non-smoker or ex-smoker (no smoking in previous 12 weeks, ≤10 pack years).
* Screening and Day -7 AM fraction of inhaled nitric oxide (FeNO) values > 40ppb. Both screening and Day -7 AM FeNO values for treatment Period 1 need to be > 40ppb for the subject to be eligible.
* Bodyweight and BMI: Bodyweight >=50 kg and body mass index (BMI) within the range 18.0 40.0 kg/m2 (inclusive)
* Male OR Female:
* Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG[ test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as:
* Pre-menopausal females reporting one of the following:

Tubal ligation Hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion Hysterectomy Bilateral Oophorectomy

* Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause [refer to laboratory reference ranges for confirmatory levels]). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until after the last dose of study medication and completion of the follow-up visit
* The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* A history of life-threatening asthma, which is defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 5 years
* Other significant pulmonary diseases to include (but not limited to): pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma.
* Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of screening that led to a change in asthma management OR in the opinion of the Investigator, is expected to affect the subject's asthma status OR the subject's ability to participate in the study. However, subjects can be rescreened to allow for an adequate time period (of at least 4 weeks) between resolution of the infection and the date of randomisation.
* Asthma Exacerbation: Any asthma exacerbation requiring oral corticosteroids within 12 weeks of screening or that resulted in overnight hospitalization requiring additional treatment for asthma within 6 months prior to screening.
* Pre-defined concomitant medications and restrictions of nitrate-rich foods
* Tobacco Use: Current smokers or a smoking history of >=10 pack years. A subject may not have used any inhaled tobacco products in 12 weeks preceding the screening visit.
* Previous Participation: Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Other concurrent Diseases/Abnormalities: A subject has any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the study results if the condition/disease exacerbated during the study.
* The list of additional excluded conditions/diseases includes, but is not limited to the following:
* Congestive heart failure-Known aortic aneurysm
* Clinically significant coronary heart disease-Clinically significant cardiac arrhythmia
* Stroke within 3 months of Visit 1-Uncontrolled hypertension
* Recent or poorly controlled peptic ulcer-Haematologic, hepatic, or renal disease
* Immunologic compromise-Current malignancy
* Tuberculosis (current or untreated)-Cushing's disease
* Addison's disease-Uncontrolled diabetes mellitus
* Liver cirrhosis-Systemic Lupus Erythematosus
* Uncontrolled thyroid disorder-Recent history of drug or alcohol abuse
* Oropharyngeal examination: A subject will not be eligible if he/she has clinical visual evidence of oral candidiasis at screening.
* Pregnancy and Lactating Females:
* Pregnant females as determined by positive serum hCG test at screening or by positive urine hCG test prior to dosing.
* Lactating females
* Allergies:
* Milk Protein Allergy: History of severe milk protein allergy.
* Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the Dry Powder Inhaler (DPI) (i.e., lactose or magnesium stearate).
* Historical Allergy: History of drug or other allergy that, in the opinion of investigator or GSK Medical Monitor, contraindicates their participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Newtown, Wellington, New Zealand

REFERENCES:
- [Derived] Daley-Yates P, Keppler B, Baines A, Bardsley G, Fingleton J. Metabolomic changes related to airway inflammation, asthma pathogenesis and systemic activity following inhaled fluticasone furoate/vilanterol: a randomized controlled trial. Respir Res. 2022 Sep 20;23(1):258. doi: 10.1186/s12931-022-02164-w. PMID 36127726
- [Derived] Bardsley G, Daley-Yates P, Baines A, Kempsford R, Williams M, Mallon T, Braithwaite I, Riddell K, Joshi S, Bareille P, Beasley R, Fingleton J; study team. Anti-inflammatory duration of action of fluticasone furoate/vilanterol trifenatate in asthma: a cross-over randomised controlled trial. Respir Res. 2018 Jul 13;19(1):133. doi: 10.1186/s12931-018-0836-6. PMID 30001712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double blind, placebo-controlled, two-period, crossover repeat dose study in adult participants with asthma. The study was conducted from 29 April 2016 to 21 February 2017, at a single site in New Zealand.
Pre-assignment Details: Total 36 participants were screened, of which 8 participants were screen failures. Of the 28 participants who were enrolled in the study, 27 participants were randomized as 1 participant withdrew before randomization. The study had Run-in period of 7 days, which was followed by a Treatment period (TP) 1, a wash-out period of 21 days and TP2.
Groups:
- Fluticasone Furoate/Vilanterol (FF/VI) Followed by Placebo: Participants were administered with FF/VI 100/25 microgram (mcg) during TP 1 followed by matching Placebo during TP 2 through a dry powder inhaler (DPI) once daily each morning for 14 days. There was a 21-day monitoring/washout period between two treatments in this two-period crossover study. Participants with any upper respiratory disorders including allergic rhinitis (both seasonal and perennial) and chronic rhinosinusitis (with or without nasal polyps), any participant who was on chronic maintenance therapies for these conditions were continued on their current standard of care medications (intranasal corticosteroids, antihistamines, cromones) throughout the entire duration of the study.
- Placebo Followed by FF/VI: Participants were administered with Placebo during TP 1 followed by FF/VI 100/25 mcg during TP 2 through DPI once daily in each morning for 14 days. There was a 21-day monitoring/washout period between two treatments in this two-period crossover study. Participants with any upper respiratory disorders including allergic rhinitis (both seasonal and perennial) and chronic rhinosinusitis (with or without nasal polyps), any participant who was on chronic maintenance therapies for these conditions were continued on their current standard of care medications (intranasal corticosteroids, antihistamines, cromones) throughout the entire duration of the study.
Period: Treatment Period 1 (35 Days)
Arm/Group | Fluticasone Furoate/Vilanterol (FF/VI) Followed by Placebo | Placebo Followed by FF/VI
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Washout Period (21 Days)
Arm/Group | Fluticasone Furoate/Vilanterol (FF/VI) Followed by Placebo | Placebo Followed by FF/VI
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Treatment Period 2 (35 Days)
Arm/Group | Fluticasone Furoate/Vilanterol (FF/VI) Followed by Placebo | Placebo Followed by FF/VI
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total (Placebo+FF/VI 100/25mcg): In this two-period crossover study, participants received FF/VI 100/25 mcg or matching placebo through DPI once daily in each morning for 14 days either in TP 1 or TP 2 as per randomization schedule. There was a 21-days monitoring/washout period between two treatments during which participants were allowed to take rescue medication if required. Participants with any upper respiratory disorders including allergic rhinitis (both seasonal and perennial) and chronic rhinosinusitis (with or without nasal polyps), any participant who was on chronic maintenance therapies for these conditions were continued on their current standard of care medications (intranasal corticosteroids, antihistamines, cromones) throughout the entire duration of the study.
Arm/Group | Total (Placebo+FF/VI 100/25mcg)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.5 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21
  Asian and White | 1
  Native Hawaiin or other Pacific Islander and White | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fraction of Exhaled Nitric Oxide (FeNO) Over Time Following the Cessation of Repeat Dose Treatment With FF/VI
Description: FeNO is non-invasive marker of airway inflammation in asthma participants. It was measured by the participants, using Niox Vero device at AM (pre-dose) and PM on Day -7 and all way through Day 29 of each TP. The FeNO measurements were done over time following stop of repeat dose treatment with FF/VI. Change from Baseline was measured as ratio of post-dose visit value to Baseline value. Baseline was defined as Day 1(Pre-dose). Subject level Baseline defined as the mean of Baseline across periods for each participant. Period level Baseline defined as the difference between the Baseline and subject level Baseline for each period and each participant. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Summary of ratio from Baseline for exhaled nitric oxide reported as Geometric mean and Geometric coefficient of Variation. NA indicates data was not available.
Time Frame: Baseline and up to Day 29 in each treatment period
Population: The Pharmacodynamic (PD) Population consisted of all the participants from the All Subject population who had at least one PD assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of exhaled Nitric Oxide
Groups:
- Placebo: Participants received matching Placebo in either of TP 1 or TP 2 through DPI once daily in each morning for 14 days. There was a 21-day monitoring/washout period between two treatments in this two-period crossover study. Participants with any upper respiratory disorders including allergic rhinitis (both seasonal and perennial) and chronic rhinosinusitis (with or without nasal polyps), any participant who was on chronic maintenance therapies for these conditions were continued on their current standard of care medications (intranasal corticosteroids, antihistamines, cromones) throughout the entire duration of the study.
- FF/VI 100/25mcg: Participants received FF/VI 100/25 mcg in either of TP 1 or TP 2 through DPI once daily in each morning for 14 days. There was a 21-day monitoring/washout period between two treatments in this two-period crossover study. Participants with any upper respiratory disorders including allergic rhinitis (both seasonal and perennial) and chronic rhinosinusitis (with or without nasal polyps), any participant who was on chronic maintenance therapies for these conditions were continued on their current standard of care medications (intranasal corticosteroids, antihistamines, cromones) throughout the entire duration of the study.
Arm/Group | Placebo | FF/VI 100/25mcg
Number analyzed (Participants) | 27 | 27
Ratio of exhaled Nitric Oxide
  Day 1, AM (n=27,27) | 1.042 (31.5499) | 0.371 (47.3672)
  Day 1, PM (n=27,27) | 0.985 (26.4785) | 0.321 (51.5233)
  Day 2, AM (n=27,27) | 1.012 (27.3017) | 0.373 (71.6824)
  Day 2, PM (n=27,27) | 0.957 (26.3328) | 0.346 (52.6225)
  Day 3, AM (n=27,27) | 0.987 (24.6102) | 0.442 (60.8203)
  Day 3, PM (n=27,27) | 0.922 (23.6705) | 0.417 (51.1903)
  Day 4, AM (n=27,27) | 1.007 (34.9235) | 0.536 (60.5532)
  Day 4, PM (n=27,27) | 0.857 (23.7972) | 0.484 (48.1593)
  Day 5, AM (n=27,27) | 0.834 (24.4572) | 0.515 (53.5926)
  Day 5, PM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 5, PM (n=26,26) | 0.734 (27.1308) | 0.473 (46.6144)
  Day 6, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 6, AM (n=26,26) | 0.794 (31.5924) | 0.525 (50.7361)
  Day 6, PM (n=24,26): number analyzed (Participants) | 24 | 26
  Day 6, PM (n=24,26) | 0.783 (30.8200) | 0.470 (43.8128)
  Day 7, AM (n=27,27) | 0.826 (31.4676) | 0.484 (49.0454)
  Day 7, PM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 7, PM (n=25,25) | 0.774 (32.7473) | 0.487 (49.9617)
  Day 8, AM (n=25,27) | 0.830 (40.7773) | 0.554 (47.5854)
  Day 8, PM (n=27,26): number analyzed (Participants) | 27 | 26
  Day 8, PM (n=27,26) | 0.834 (30.4030) | 0.545 (42.1101)
  Day 9, AM (n=27,27) | 0.935 (35.7583) | 0.594 (45.0429)
  Day 9, PM (n=27,27) | 0.924 (32.1314) | 0.607 (46.3872)
  Day 10, AM (n=24,26): number analyzed (Participants) | 24 | 26
  Day 10, AM (n=24,26) | 1.022 (34.4740) | 0.658 (41.3710)
  Day 10, PM (n=27,27) | 0.989 (35.1066) | 0.660 (41.4832)
  Day 11, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 11, AM (n=26,26) | 1.092 (37.7142) | 0.756 (40.9942)
  Day 11, PM (n=27,27) | 1.029 (28.6618) | 0.723 (45.9281)
  Day 12, AM (n=27,27) | 1.028 (29.9667) | 0.717 (42.8654)
  Day 12, PM (n=27,27) | 1.004 (28.5673) | 0.691 (43.1839)
  Day 13, AM (n=27,25): number analyzed (Participants) | 27 | 25
  Day 13, AM (n=27,25) | 1.068 (34.0090) | 0.744 (38.4939)
  Day 13, PM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 13, PM (n=25,25) | 0.955 (40.2945) | 0.739 (39.5506)
  Day 14, AM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 14, AM (n=26,27) | 1.008 (45.5319) | 0.770 (43.7613)
  Day 14, PM (n=25,26): number analyzed (Participants) | 25 | 26
  Day 14, PM (n=25,26) | 0.955 (45.5768) | 0.634 (76.0516)
  Day 15, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 15, AM (n=26,26) | 0.977 (51.5523) | 0.731 (40.4602)
  Day 15, PM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 15, PM (n=25,25) | 0.940 (42.3660) | 0.700 (48.1949)
  Day 16, AM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 16, AM (n=26,27) | 1.029 (51.1876) | 0.727 (44.7703)
  Day 16, PM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 16, PM (n=26,27) | 1.019 (38.1690) | 0.718 (50.7656)
  Day 17, AM (n=25,26): number analyzed (Participants) | 25 | 26
  Day 17, AM (n=25,26) | 1.049 (40.1495) | 0.770 (44.3320)
  Day 17, PM (n=18,16): number analyzed (Participants) | 18 | 16
  Day 17, PM (n=18,16) | 0.967 (38.4731) | 0.765 (59.4286)
  Day 18, AM (n=17,14): number analyzed (Participants) | 17 | 14
  Day 18, AM (n=17,14) | 0.935 (39.0474) | 0.724 (54.2082)
  Day 18, PM (n=14,10): number analyzed (Participants) | 14 | 10
  Day 18, PM (n=14,10) | 0.926 (39.2470) | 0.619 (58.6249)
  Day 19, AM (n=14,10): number analyzed (Participants) | 14 | 10
  Day 19, AM (n=14,10) | 1.015 (42.2250) | 0.722 (51.2962)
  Day 19, PM (n=12,6): number analyzed (Participants) | 12 | 6
  Day 19, PM (n=12,6) | 0.911 (30.6911) | 0.571 (48.1910)
  Day 20, AM (n=12,6): number analyzed (Participants) | 12 | 6
  Day 20, AM (n=12,6) | 0.958 (43.0056) | 0.667 (45.5449)
  Day 20, PM (n=7,5): number analyzed (Participants) | 7 | 5
  Day 20, PM (n=7,5) | 0.828 (39.6562) | 0.588 (54.7676)
  Day 21, AM (n=7,6): number analyzed (Participants) | 7 | 6
  Day 21, AM (n=7,6) | 0.892 (35.8531) | 0.743 (54.8750)
  Day 21, PM (n=7,5): number analyzed (Participants) | 7 | 5
  Day 21, PM (n=7,5) | 0.934 (40.4076) | 0.637 (63.2223)
  Day 22, AM (n=6,5): number analyzed (Participants) | 6 | 5
  Day 22, AM (n=6,5) | 0.845 (45.8754) | 0.705 (82.0353)
  Day 22, PM (n=6,5): number analyzed (Participants) | 6 | 5
  Day 22, PM (n=6,5) | 0.822 (43.0801) | 0.622 (75.8988)
  Day 23, AM (n=7,5): number analyzed (Participants) | 7 | 5
  Day 23, AM (n=7,5) | 0.925 (51.4896) | 0.749 (76.0176)
  Day 23, PM (n=2,1): number analyzed (Participants) | 2 | 1
  Day 23, PM (n=2,1) | 0.898 (116.9108) | 1.000 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 24, AM (n=2,1): number analyzed (Participants) | 2 | 1
  Day 24, AM (n=2,1) | 0.914 (130.0375) | 1.144 (NA) — Standard deviation could not be computed as a single participant was analyzed.
  Day 24, PM (n=1,1): number analyzed (Participants) | 1 | 1
  Day 24, PM (n=1,1) | 0.671 (NA) — Standard deviation could not be computed as a single participant was analyzed | 0.911 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 25, AM (n=1,0): number analyzed (Participants) | 1 | 0
  Day 25, AM (n=1,0) | 0.548 (NA) — Standard deviation could not be computed as a single participant was analyzed |
  Day 26, PM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 26, PM (n=0,1) |  | 0.989 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 28, AM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 28, AM (n=0,1) |  | 1.044 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 28, PM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 28, PM (n=0,1) |  | 0.767 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 29, AM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 29, AM (n=0,1) |  | 0.911 (NA) — Standard deviation could not be computed as a single participant was analyzed
Statistical Analysis 1: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.36, 95% CI 2-sided [0.31 to 0.43] — Ratio of FF/VI 100/25mcg versus (Vs) Placebo for Day 1, AM
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.33, 95% CI 2-sided [0.28 to 0.39] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 1, PM
Statistical Analysis 3: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.38, 95% CI 2-sided [0.32 to 0.45] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 2, AM
Statistical Analysis 4: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.37, 95% CI 2-sided [0.31 to 0.44] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 2, PM
Statistical Analysis 5: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.46, 95% CI 2-sided [0.39 to 0.54] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 3, AM
Statistical Analysis 6: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.47, 95% CI 2-sided [0.40 to 0.56] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 3, PM
Statistical Analysis 7: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.56, 95% CI 2-sided [0.47 to 0.66] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 4, AM
Statistical Analysis 8: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.58, 95% CI 2-sided [0.49 to 0.69] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 4, PM
Statistical Analysis 9: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.63, 95% CI 2-sided [0.53 to 0.75] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 5, AM
Statistical Analysis 10: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.67, 95% CI 2-sided [0.57 to 0.80] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 5, PM
Statistical Analysis 11: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.67, 95% CI 2-sided [0.56 to 0.80] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 6, AM
Statistical Analysis 12: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.62, 95% CI 2-sided [0.52 to 0.74] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 6, PM
Statistical Analysis 13: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.60, 95% CI 2-sided [0.51 to 0.71] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 7, AM
Statistical Analysis 14: Comparison: Placebo vs FF/VI 100/25mcg; Ratio of FF/VI 100/25mcg Vs Placebo for Day 8, AM; Test type: Other; Ratio = 0.62, 95% CI 2-sided [0.52 to 0.74] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 7, PM
Statistical Analysis 15: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.69, 95% CI 2-sided [0.58 to 0.81] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 8, AM
Statistical Analysis 16: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.68, 95% CI 2-sided [0.57 to 0.80] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 8, PM
Statistical Analysis 17: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.66, 95% CI 2-sided [0.56 to 0.78] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 9, AM
Statistical Analysis 18: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.68, 95% CI 2-sided [0.57 to 0.80] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 9, PM
Statistical Analysis 19: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.66, 95% CI 2-sided [0.55 to 0.78] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 10, AM
Statistical Analysis 20: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.68, 95% CI 2-sided [0.58 to 0.81] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 10, PM
Statistical Analysis 21: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.73, 95% CI 2-sided [0.61 to 0.86] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 11, AM
Statistical Analysis 22: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.73, 95% CI 2-sided [0.61 to 0.86] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 11, PM
Statistical Analysis 23: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.72, 95% CI 2-sided [0.61 to 0.85] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 12, AM
Statistical Analysis 24: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.71, 95% CI 2-sided [0.60 to 0.84] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 12, PM
Statistical Analysis 25: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.72, 95% CI 2-sided [0.61 to 0.86] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 13, AM
Statistical Analysis 26: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.78, 95% CI 2-sided [0.66 to 0.93] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 13, PM
Statistical Analysis 27: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.79, 95% CI 2-sided [0.66 to 0.93] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 14, AM
Statistical Analysis 28: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.67, 95% CI 2-sided [0.56 to 0.79] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 14, PM
Statistical Analysis 29: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.79, 95% CI 2-sided [0.66 to 0.93] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 15, AM
Statistical Analysis 30: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.79, 95% CI 2-sided [0.66 to 0.94] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 15, PM
Statistical Analysis 31: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.74, 95% CI 2-sided [0.62 to 0.87] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 16, AM
Statistical Analysis 32: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.73, 95% CI 2-sided [0.61 to 0.86] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 16, PM
Statistical Analysis 33: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.77, 95% CI 2-sided [0.65 to 0.91] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 17, AM
Statistical Analysis 34: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.81, 95% CI 2-sided [0.65 to 1.01] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 17, PM
Statistical Analysis 35: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.77, 95% CI 2-sided [0.61 to 0.96] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 18, AM
Statistical Analysis 36: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.77, 95% CI 2-sided [0.59 to 1.00] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 18, PM
Statistical Analysis 37: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.81, 95% CI 2-sided [0.63 to 1.05] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 19, AM
Statistical Analysis 38: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.72, 95% CI 2-sided [0.52 to 1.00] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 19, PM
Statistical Analysis 39: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.78, 95% CI 2-sided [0.56 to 1.09] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 20, AM
Statistical Analysis 40: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.78, 95% CI 2-sided [0.53 to 1.14] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 20, PM
Statistical Analysis 41: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.85, 95% CI 2-sided [0.59 to 1.22] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 21, AM
Statistical Analysis 42: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.75, 95% CI 2-sided [0.50 to 1.13] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 21, PM
Statistical Analysis 43: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.83, 95% CI 2-sided [0.55 to 1.25] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 22, AM
Statistical Analysis 44: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.77, 95% CI 2-sided [0.51 to 1.16] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 22, PM
Statistical Analysis 45: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.99, 95% CI 2-sided [0.66 to 1.49] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 23, AM
Statistical Analysis 46: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.67, 95% CI 2-sided [0.29 to 1.51] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 23, PM
Statistical Analysis 47: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Ratio = 0.72, 95% CI 2-sided [0.32 to 1.64] — Ratio of FF/VI 100/25mcg Vs Placebo for Day 24, AM

2. Secondary Outcome: Change From Baseline in FeNO Over the FF/VI Treatment Period
Description: In participants with asthma the FeNO is a non-invasive marker of airway inflammation. The FeNO was measured by the participants AM (pre-dose) and PM on Day -7 and all the way through Day 29 of each treatment period. The measurements were recorded using Niox Vero device provided at the site. These FeNO measurements were done throughout the treatment period. Change from Baseline was measured by the value at post-dose visit minus the Baseline value. Baseline was defined as Day 1(Pre-dose). Subject level Baseline is defined as the mean of Baseline across periods for each participant. Period level Baseline is defined as the difference between the Baseline and subject level Baseline for each period and each participant. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data was not available.
Time Frame: Baseline and up to Day 29 in each treatment period
Population: PD Population.
Measure: Mean (Standard Deviation); unit: Parts per billion
Arm/Group | Placebo | FF/VI 100/25mcg
Number analyzed (Participants) | 27 | 27
Parts per billion
  Day 1, AM (n=27,27) | 1.9 (24.39) | -63.3 (45.47)
  Day 1, PM (n=27,27) | -0.5 (24.55) | -68.5 (49.07)
  Day 2, AM (n=27,27) | 1.3 (27.67) | -63.5 (53.63)
  Day 2, PM (n=27,27) | -3.1 (24.64) | -66.1 (48.26)
  Day 3, AM (n=27,27) | -0.8 (25.07) | -56.6 (53.97)
  Day 3, PM (n=27,27) | -7.9 (21.18) | -59.8 (47.32)
  Day 4, AM (n=27,27) | 1.2 (33.27) | -48.6 (50.54)
  Day 4, PM (n=27,27) | -11.6 (17.93) | -51.5 (42.12)
  Day 5, AM (n=27,27) | -15.3 (22.49) | -48.9 (47.09)
  Day 5, PM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 5, PM (n=26,26) | -22.1 (19.45) | -54.0 (45.00)
  Day 6, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 6, AM (n=26,26) | -17.6 (24.37) | -47.1 (42.19)
  Day 6, PM (n=24,26): number analyzed (Participants) | 24 | 26
  Day 6, PM (n=24,26) | -19.4 (25.76) | -54.0 (43.96)
  Day 7, AM (n=27,27) | -15.4 (24.26) | -50.0 (43.19)
  Day 7, PM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 7, PM (n=25,25) | -19.9 (25.92) | -46.4 (42.73)
  Day 8, AM (n=25,27): number analyzed (Participants) | 25 | 27
  Day 8, AM (n=25,27) | -14.2 (30.00) | -42.7 (44.14)
  Day 8, PM (n=27,26): number analyzed (Participants) | 27 | 26
  Day 8, PM (n=27,26) | -15.3 (24.70) | -46.1 (40.39)
  Day 9, AM (n=27,27) | -5.7 (29.23) | -40.1 (37.45)
  Day 9, PM (n=27,27) | -5.3 (23.53) | -38.7 (40.36)
  Day 10, AM (n=24,26) | 4.1 (27.86) | -31.6 (31.50)
  Day 10, PM (n=27,27) | 3.8 (28.99) | -32.8 (37.47)
  Day 11, AM (n=26,26) | 12.8 (31.82) | -23.8 (39.65)
  Day 11, PM (n=27,27) | 6.2 (34.03) | -26.4 (41.33)
  Day 12, AM (n=27,27) | 3.1 (24.79) | -25.7 (36.64)
  Day 12, PM (n=27,27) | 1.3 (25.08) | -29.4 (37.19)
  Day 13, AM (n=27,25): number analyzed (Participants) | 27 | 25
  Day 13, AM (n=27,25) | 8.3 (35.47) | -23.3 (30.09)
  Day 13, PM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 13, PM (n=25,25) | -1.6 (38.12) | -26.2 (39.97)
  Day 14, AM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 14, AM (n=26,27) | 4.7 (45.42) | -23.5 (38.84)
  Day 14, PM (n=25,26): number analyzed (Participants) | 25 | 26
  Day 14, PM (n=25,26) | -3.4 (42.26) | -30.9 (43.69)
  Day 15, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 15, AM (n=26,26) | -1.6 (47.88) | -25.8 (37.76)
  Day 15, PM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 15, PM (n=25,25) | -3.7 (49.33) | -27.9 (43.14)
  Day 16, AM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 16, AM (n=26,27) | 3.7 (48.00) | -26.7 (43.16)
  Day 16, PM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 16, PM (n=26,27) | 4.5 (37.40) | -26.6 (43.37)
  Day 17, AM (n=25,26): number analyzed (Participants) | 25 | 26
  Day 17, AM (n=25,26) | 6.1 (42.81) | -20.9 (39.31)
  Day 17, PM (n=18,16): number analyzed (Participants) | 18 | 16
  Day 17, PM (n=18,16) | -8.5 (29.54) | -19.6 (48.58)
  Day 18, AM (n=17,14): number analyzed (Participants) | 17 | 14
  Day 18, AM (n=17,14) | -7.5 (32.10) | -27.3 (44.36)
  Day 18, PM (n=14,10): number analyzed (Participants) | 14 | 10
  Day 18, PM (n=14,10) | -6.2 (23.93) | -38.3 (42.90)
  Day 19, AM (n=14,10): number analyzed (Participants) | 14 | 10
  Day 19, AM (n=14,10) | -2.8 (27.47) | -30.7 (50.03)
  Day 19, PM (n=12,6): number analyzed (Participants) | 12 | 6
  Day 19, PM (n=12,6) | -9.3 (24.19) | -52.2 (49.82)
  Day 20, AM (n=12,6): number analyzed (Participants) | 12 | 6
  Day 20, AM (n=12,6) | 0.1 (27.71) | -40.2 (46.27)
  Day 20, PM (n=7,5): number analyzed (Participants) | 7 | 5
  Day 20, PM (n=7,5) | -8.7 (21.68) | -59.0 (63.82)
  Day 21, AM (n=7,6): number analyzed (Participants) | 7 | 6
  Day 21, AM (n=7,6) | -6.6 (24.08) | -32.7 (56.23)
  Day 21, PM (n=7,5): number analyzed (Participants) | 7 | 5
  Day 21, PM (n=7,5) | -3.0 (25.83) | -51.2 (58.37)
  Day 22, AM (n=6,5): number analyzed (Participants) | 6 | 5
  Day 22, AM (n=6,5) | -7.5 (27.54) | -37.0 (66.25)
  Day 22, PM (n=6,5): number analyzed (Participants) | 6 | 5
  Day 22, PM (n=6,5) | -11.5 (27.52) | -51.8 (63.96)
  Day 23, AM (n=7,5): number analyzed (Participants) | 7 | 5
  Day 23, AM (n=7,5) | -0.6 (29.53) | -37.0 (71.04)
  Day 23, PM (n=2,1): number analyzed (Participants) | 2 | 1
  Day 23, PM (n=2,1) | -0.5 (54.45) | 0.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.
  Day 24, AM (n=2,1): number analyzed (Participants) | 2 | 1
  Day 24, AM (n=2,1) | 2.0 (59.40) | 13.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.
  Day 24, PM (n=1,1): number analyzed (Participants) | 1 | 1
  Day 24, PM (n=1,1) | -24.0 (NA) — Standard deviation could not be computed as a single participant was analyzed. | -8.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.
  Day 25, AM (n=1,0): number analyzed (Participants) | 1 | 0
  Day 25, AM (n=1,0) | -33.0 (NA) — Standard deviation could not be computed as a single participant was analyzed. |
  Day 26, PM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 26, PM (n=0,1) |  | -1.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.
  Day 28, AM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 28, AM (n=0,1) |  | 4.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.
  Day 28, PM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 28, PM (n=0,1) |  | -21.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.
  Day 29, AM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 29, AM (n=0,1) |  | -8.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.

3. Secondary Outcome: Change From Baseline in Peak Expiratory Flow (PEF) During Treatment and Following Cessation of Repeat Dose Treatment With FF/VI
Description: The PEF is a lung function evaluation assessed using a PEF meter. It was defined as the maximum amount of air exhaled during forced exhalation with lungs fully inflated. For PEF measurements the best of the 3 recordings were recorded AM and PM (i.e every 12 hours), from Day-7 through to Day 29 of TP1, and then from Day 1 of TP2 through to the (29). Change from Baseline was measured by the value at post-dose visit minus the Baseline value. Baseline was defined as Day 1(Pre-dose). Subject level Baseline is defined as the mean of Baseline across periods for each participant. Period level Baseline is defined as the difference between the Baseline and subject level Baseline for each period and each participant. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data was not available.
Time Frame: Baseline and up to Day 29 in TP1; Baseline and up to follow up (Day 29) in TP2
Population: PD population.
Measure: Mean (Standard Deviation); unit: Liter per minute
Arm/Group | Placebo | FF/VI 100/25mcg
Number analyzed (Participants) | 27 | 27
Liter per minute
  Day 1, AM (n=27,27) | -1.0 (67.11) | 44.6 (55.54)
  Day 1, PM (n=27,27) | 17.4 (69.59) | 54.5 (63.23)
  Day 2, AM (n=27,27) | 5.1 (61.50) | 32.4 (55.35)
  Day 2, PM (n=27,27) | 16.6 (74.02) | 37.2 (53.42)
  Day 3, AM (n=27,27) | 9.0 (58.49) | 24.3 (58.56)
  Day 3, PM (n=27,27) | 20.4 (69.10) | 47.3 (52.80)
  Day 4, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 4, AM (n=26,26) | 18.3 (61.63) | 28.8 (54.42)
  Day 4, PM (n=27,27) | 36.0 (85.62) | 43.9 (56.01)
  Day 5, AM (n=27,26): number analyzed (Participants) | 27 | 26
  Day 5, AM (n=27,26) | 19.7 (61.28) | 25.4 (49.86)
  Day 5, PM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 5, PM (n=26,27) | 21.5 (75.94) | 30.9 (49.67)
  Day 6, AM (n=25,26): number analyzed (Participants) | 25 | 26
  Day 6, AM (n=25,26) | -0.4 (69.89) | 4.1 (61.63)
  Day 6, PM (n=24,26): number analyzed (Participants) | 24 | 26
  Day 6, PM (n=24,26) | 11.3 (75.26) | 28.5 (52.75)
  Day 7, AM (n=27,27) | 11.5 (71.97) | 17.0 (55.89)
  Day 7, PM (n=24,26): number analyzed (Participants) | 24 | 26
  Day 7, PM (n=24,26) | 11.8 (75.33) | 21.8 (55.70)
  Day 8, AM (n=27,27) | -1.6 (73.80) | 2.6 (51.94)
  Day 8, PM (n=27,27) | 13.1 (61.79) | 9.1 (56.68)
  Day 9, AM (n=27,26): number analyzed (Participants) | 27 | 26
  Day 9, AM (n=27,26) | -7.2 (80.69) | -14.7 (74.06)
  Day 9, PM (n=27,27) | 9.1 (73.71) | -1.7 (58.12)
  Day 10, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 10, AM (n=26,26) | -19.6 (76.63) | -19.9 (68.55)
  Day 10, PM (n=27,26): number analyzed (Participants) | 27 | 26
  Day 10, PM (n=27,26) | -1.7 (84.64) | 12.6 (52.16)
  Day 11, AM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 11, AM (n=26,27) | -12.8 (74.84) | -12.3 (56.24)
  Day 11, PM (n=27,27) | 15.8 (76.76) | -7.3 (63.12)
  Day 12, AM (n=24,26): number analyzed (Participants) | 24 | 26
  Day 12, AM (n=24,26) | -11.0 (83.14) | -23.5 (64.35)
  Day 12, PM (n=26,27): number analyzed (Participants) | 26 | 27
  Day 12, PM (n=26,27) | -2.4 (71.17) | -5.9 (66.19)
  Day 13, AM (n=27,26): number analyzed (Participants) | 27 | 26
  Day 13, AM (n=27,26) | -20.6 (77.50) | -35.1 (67.19)
  Day 13, PM (n=25,26): number analyzed (Participants) | 25 | 26
  Day 13, PM (n=25,26) | 17.0 (104.76) | -13.0 (61.78)
  Day 14, AM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 14, AM (n=25,25) | -31.5 (77.48) | -13.6 (65.25)
  Day 14, PM (n=25,27): number analyzed (Participants) | 25 | 27
  Day 14, PM (n=25,27) | -0.8 (76.69) | -1.6 (58.26)
  Day 15, AM (n=25,27): number analyzed (Participants) | 25 | 27
  Day 15, AM (n=25,27) | -17.4 (59.88) | -20.4 (58.86)
  Day 15, PM (n=25,25): number analyzed (Participants) | 25 | 25
  Day 15, PM (n=25,25) | -15.0 (67.65) | -7.8 (64.72)
  Day 16, AM (n=25,26): number analyzed (Participants) | 25 | 26
  Day 16, AM (n=25,26) | -27.0 (66.70) | -30.2 (75.78)
  Day 16, PM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 16, PM (n=26,26) | -8.1 (74.86) | 0.7 (60.72)
  Day 17, AM (n=26,26): number analyzed (Participants) | 26 | 26
  Day 17, AM (n=26,26) | -23.4 (73.32) | -4.7 (65.85)
  Day 17, PM (n=18,16): number analyzed (Participants) | 18 | 16
  Day 17, PM (n=18,16) | 10.6 (86.60) | 8.7 (62.33)
  Day 18, AM (n=17,14): number analyzed (Participants) | 17 | 14
  Day 18, AM (n=17,14) | -14.2 (79.96) | 3.8 (71.50)
  Day 18, PM (n=14,10): number analyzed (Participants) | 14 | 10
  Day 18, PM (n=14,10) | -8.9 (90.25) | 29.6 (64.62)
  Day 19, AM (n=14,10): number analyzed (Participants) | 14 | 10
  Day 19, AM (n=14,10) | -11.4 (91.61) | -0.1 (70.24)
  Day 19, PM (n=12,6): number analyzed (Participants) | 12 | 6
  Day 19, PM (n=12,6) | 2.3 (102.76) | 27.7 (61.49)
  Day 20, AM (n=12,6): number analyzed (Participants) | 12 | 6
  Day 20, AM (n=12,6) | -8.5 (81.09) | -10.5 (71.92)
  Day 20, PM (n=7,5): number analyzed (Participants) | 7 | 5
  Day 20, PM (n=7,5) | -27.7 (46.03) | 26.6 (49.22)
  Day 21, AM (n=7,6): number analyzed (Participants) | 7 | 6
  Day 21, AM (n=7,6) | -43.3 (56.85) | 17.8 (78.20)
  Day 21, PM (n=6,4): number analyzed (Participants) | 6 | 4
  Day 21, PM (n=6,4) | -16.7 (73.86) | -19.8 (32.62)
  Day 22, AM (n=5,5): number analyzed (Participants) | 5 | 5
  Day 22, AM (n=5,5) | -48.4 (40.28) | -11.0 (103.22)
  Day 22, PM (n=6,5): number analyzed (Participants) | 6 | 5
  Day 22, PM (n=6,5) | -56.8 (46.23) | -2.0 (91.29)
  Day 23, AM (n=6,5): number analyzed (Participants) | 6 | 5
  Day 23, AM (n=6,5) | -15.0 (50.62) | 11.4 (53.62)
  Day 23, PM (n=2,1): number analyzed (Participants) | 2 | 1
  Day 23, PM (n=2,1) | -53.0 (1.41) | 1.0 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 24, AM (n=2,1): number analyzed (Participants) | 2 | 1
  Day 24, AM (n=2,1) | -23.0 (25.46) | 74.0 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 24, PM (n=1,1): number analyzed (Participants) | 1 | 1
  Day 24, PM (n=1,1) | -50.0 (NA) — Standard deviation could not be computed as a single participant was analyzed | 15.0 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 25, AM (n=1,0): number analyzed (Participants) | 1 | 0
  Day 25, AM (n=1,0) | -31.0 (NA) — Standard deviation could not be computed as a single participant was analyzed |
  Day 26, PM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 26, PM (n=0,1) |  | -62.0 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 27, AM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 27, AM (n=0,1) |  | 82.0 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 28, AM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 28, AM (n=0,1) |  | -42.0 (NA) — Standard deviation could not be computed as a single participant was analyzed
  Day 29, AM (n=0,1): number analyzed (Participants) | 0 | 1
  Day 29, AM (n=0,1) |  | 6.0 (NA) — Standard deviation could not be computed as a single participant was analyzed.
Statistical Analysis 1: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 45.86, 95% CI 2-sided [23.69 to 68.03] — Difference of FF/VI 100/25mcg Vs Placebo for Day 1, AM
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 45.37, 95% CI 2-sided [23.20 to 67.55] — Difference of FF/VI 100/25mcg Vs Placebo for Day 1, PM
Statistical Analysis 3: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 34.03, 95% CI 2-sided [11.86 to 56.21] — Difference of FF/VI 100/25mcg Vs Placebo for Day 2, AM
Statistical Analysis 4: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 31.56, 95% CI 2-sided [9.38 to 53.73] — Difference of FF/VI 100/25mcg Vs Placebo for Day 2, PM
Statistical Analysis 5: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 22.86, 95% CI 2-sided [0.68 to 45.03] — Difference of FF/VI 100/25mcg Vs Placebo for Day 3, AM
Statistical Analysis 6: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 36.94, 95% CI 2-sided [14.77 to 59.12] — Difference of FF/VI 100/25mcg Vs Placebo for Day 3, PM
Statistical Analysis 7: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 19.33, 95% CI 2-sided [-3.00 to 41.66] — Difference of FF/VI 100/25mcg Vs Placebo for Day 4, AM
Statistical Analysis 8: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 20.85, 95% CI 2-sided [-1.32 to 43.03] — Difference of FF/VI 100/25mcg Vs Placebo for Day 4, PM
Statistical Analysis 9: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 16.82, 95% CI 2-sided [-5.47 to 39.11] — Difference of FF/VI 100/25mcg Vs Placebo for Day 5, AM
Statistical Analysis 10: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 21.86, 95% CI 2-sided [-0.41 to 44.14] — Difference of FF/VI 100/25mcg Vs Placebo for Day 5, PM
Statistical Analysis 11: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 13.05, 95% CI 2-sided [-9.57 to 35.67] — Difference of FF/VI 100/25mcg Vs Placebo for Day 6, AM
Statistical Analysis 12: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 28.68, 95% CI 2-sided [5.38 to 51.98] — Difference of FF/VI 100/25mcg Vs Placebo for Day 6, PM
Statistical Analysis 13: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 17.09, 95% CI 2-sided [-5.08 to 39.26] — Difference of FF/VI 100/25mcg Vs Placebo for Day 7, AM
Statistical Analysis 14: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 23.61, 95% CI 2-sided [0.28 to 46.94] — Difference of FF/VI 100/25mcg Vs Placebo for Day 7, PM
Statistical Analysis 15: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 12.87, 95% CI 2-sided [-9.30 to 35.05] — Difference of FF/VI 100/25mcg Vs Placebo for Day 8, AM
Statistical Analysis 16: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 7.50, 95% CI 2-sided [-14.67 to 29.68] — Difference of FF/VI 100/25mcg Vs Placebo for Day 8, PM
Statistical Analysis 17: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 3.32, 95% CI 2-sided [-19.11 to 25.74] — Difference of FF/VI 100/25mcg Vs Placebo for Day 9, AM
Statistical Analysis 18: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 3.83, 95% CI 2-sided [-18.34 to 26.00] — Difference of FF/VI 100/25mcg Vs Placebo for Day 9, PM
Statistical Analysis 19: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 11.36, 95% CI 2-sided [-11.11 to 33.82] — Difference of FF/VI 100/25mcg Vs Placebo for Day 10, AM
Statistical Analysis 20: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 27.73, 95% CI 2-sided [5.43 to 50.03] — Difference of FF/VI 100/25mcg Vs Placebo for Day 10, PM
Statistical Analysis 21: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 14.71, 95% CI 2-sided [-7.57 to 36.98] — Difference of FF/VI 100/25mcg Vs Placebo for Day 11, AM
Statistical Analysis 22: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = -6.62, 95% CI 2-sided [-28.80 to 15.55] — Difference of FF/VI 100/25mcg Vs Placebo for Day 11, PM
Statistical Analysis 23: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 4.36, 95% CI 2-sided [-18.39 to 27.11] — Difference of FF/VI 100/25mcg Vs Placebo for Day 12, AM
Statistical Analysis 24: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 8.29, 95% CI 2-sided [-13.99 to 30.57] — Difference of FF/VI 100/25mcg Vs Placebo for Day 12, PM
Statistical Analysis 25: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.64, 95% CI 2-sided [-21.64 to 22.92] — Difference of FF/VI 100/25mcg Vs Placebo for Day 13, AM
Statistical Analysis 26: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = -6.88, 95% CI 2-sided [-29.96 to 16.19] — Difference of FF/VI 100/25mcg Vs Placebo for Day 13, PM
Statistical Analysis 27: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 28.45, 95% CI 2-sided [5.76 to 51.13] — Difference of FF/VI 100/25mcg Vs Placebo for Day 14, AM
Statistical Analysis 28: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 12.31, 95% CI 2-sided [-10.13 to 34.74] — Difference of FF/VI 100/25mcg Vs Placebo for Day 14, PM
Statistical Analysis 29: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 4.10, 95% CI 2-sided [-18.16 to 26.36] — Difference of FF/VI 100/25mcg Vs Placebo for Day 15, AM
Statistical Analysis 30: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 18.87, 95% CI 2-sided [-3.89 to 41.63] — Difference of FF/VI 100/25mcg Vs Placebo for Day 15, PM
Statistical Analysis 31: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 6.35, 95% CI 2-sided [-16.17 to 28.88] — Difference of FF/VI 100/25mcg Vs Placebo for Day 16, AM
Statistical Analysis 32: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 19.07, 95% CI 2-sided [-3.27 to 41.41] — Difference of FF/VI 100/25mcg Vs Placebo for Day 16, PM
Statistical Analysis 33: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 29.51, 95% CI 2-sided [6.87 to 52.15] — Difference of FF/VI 100/25mcg Vs Placebo for Day 17, AM
Statistical Analysis 34: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 9.64, 95% CI 2-sided [-17.91 to 37.19] — Difference of FF/VI 100/25mcg Vs Placebo for Day 17, PM
Statistical Analysis 35: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 24.77, 95% CI 2-sided [-4.20 to 53.73] — Difference of FF/VI 100/25mcg Vs Placebo for Day 18, AM
Statistical Analysis 36: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 47.04, 95% CI 2-sided [14.63 to 79.45] — Difference of FF/VI 100/25mcg Vs Placebo for Day 18, PM
Statistical Analysis 37: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 20.11, 95% CI 2-sided [-12.30 to 52.52] — Difference of FF/VI 100/25mcg Vs Placebo for Day 19, AM
Statistical Analysis 38: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 25.13, 95% CI 2-sided [-15.02 to 65.27] — Difference of FF/VI 100/25mcg Vs Placebo for Day 19, PM
Statistical Analysis 39: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = -7.89, 95% CI 2-sided [-48.04 to 32.25] — Difference of FF/VI 100/25mcg Vs Placebo for Day 20, AM
Statistical Analysis 40: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 8.51, 95% CI 2-sided [-37.22 to 54.25] — Difference of FF/VI 100/25mcg Vs Placebo for Day 20, PM
Statistical Analysis 41: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 15.08, 95% CI 2-sided [-28.50 to 58.67] — Difference of FF/VI 100/25mcg Vs Placebo for Day 21, AM
Statistical Analysis 42: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 5.19, 95% CI 2-sided [-45.35 to 55.73] — Difference of FF/VI 100/25mcg Vs Placebo for Day 21, PM

4. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Pre-treatment and for up to 7 Days After Cessation of Repeat Dose Treatment With FF/VI
Description: FEV1 is defined as the maximal amount of air which can be exhaled forcefully in one second. Three technically acceptable FEV1 measurements were made using a spirometer, and were measured on pre-dose on Day 1, taken pre-dose on Day 14 and every morning and evening until Day 19, and in the morning on Day 21. Change from Baseline was measured by the value at post-dose visit minus the Baseline value. Baseline was defined as Day 1(Pre-dose). Subject level Baseline is defined as the mean of Baseline across periods for each participant. Period level Baseline is defined as the difference between the Baseline and subject level Baseline for each period and each participant.
Time Frame: Baseline every morning and evening until Day 21 of each treatment period
Population: PD Population
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | FF/VI 100/25mcg
Number analyzed (Participants) | 27 | 27
Liter
  Day 1, AM | 0.036 (0.4169) | 0.361 (0.3135)
  Day 1, PM | 0.180 (0.3105) | 0.383 (0.3151)
  Day 2, AM | 0.073 (0.3953) | 0.331 (0.2739)
  Day 2,PM | 0.200 (0.3902) | 0.369 (0.3166)
  Day 3,AM | 0.084 (0.3668) | 0.271 (0.2967)
  Day 3,PM | 0.213 (0.3840) | 0.319 (0.3256)
  Day 4, AM | 0.092 (0.3870) | 0.241 (0.2913)
  Day 4, PM | 0.221 (0.4187) | 0.301 (0.3163)
  Day 5, AM | 0.197 (0.3375) | 0.207 (0.2498)
  Day 7, AM | 0.124 (0.3753) | 0.102 (0.3317)
  Day 21, AM | 0.082 (0.3210) | 0.004 (0.2670)
Statistical Analysis 1: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.36, 95% CI 2-sided [0.26 to 0.46] — Difference of FF/VI 100/25mcg Vs Placebo for Day 1, AM
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.26, 95% CI 2-sided [0.16 to 0.36] — Difference of FF/VI 100/25mcg Vs Placebo for Day 1, PM
Statistical Analysis 3: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.34, 95% CI 2-sided [0.24 to 0.44] — Difference of FF/VI 100/25mcg Vs Placebo for Day 2, AM
Statistical Analysis 4: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.24, 95% CI 2-sided [0.14 to 0.34] — Difference of FF/VI 100/25mcg Vs Placebo for Day 2, PM
Statistical Analysis 5: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.26, 95% CI 2-sided [0.16 to 0.36] — Difference of FF/VI 100/25mcg Vs Placebo for Day 3, AM
Statistical Analysis 6: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.18, 95% CI 2-sided [0.08 to 0.28] — Difference of FF/VI 100/25mcg Vs Placebo for Day 3, PM
Statistical Analysis 7: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.24, 95% CI 2-sided [0.14 to 0.34] — Difference of FF/VI 100/25mcg Vs Placebo for Day 4, AM
Statistical Analysis 8: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.17, 95% CI 2-sided [0.07 to 0.27] — Difference of FF/VI 100/25mcg Vs Placebo for Day 4, PM
Statistical Analysis 9: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.03 to 0.17] — Difference of FF/VI 100/25mcg Vs Placebo for Day 5, AM
Statistical Analysis 10: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.06 to 0.14] — Difference of FF/VI 100/25mcg Vs Placebo for Day 7, AM
Statistical Analysis 11: Comparison: Placebo vs FF/VI 100/25mcg; Test type: Other; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.07 to 0.13] — Difference of FF/VI 100/25mcg Vs Placebo for Day 21, AM

ADVERSE EVENTS:
Time Frame: All the Serious adverse events (SAEs) and Adverse events (AEs) from Day 1 to upto Day 35 in each period (Total 70 days)
Description: The 'All Subjects' population comprised of all participants randomized to the treatment who received at least one dose of study treatment, was used to assess the AEs and SAEs.
Arm/Group | Placebo | FF/VI 100/25mcg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 10/27 | 14/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | FF/VI 100/25mcg (N=27)
Viral upper respiratory tract infection (Infections and infestations) | 5 | 7
Orchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT02712047/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT02712047/SAP_001.pdf